CLINICAL TRIAL: NCT05204238
Title: Follow Up of acuTe Heart failUre: a pRospective Echocardiographic and Clinical Study (FUTURE)
Acronym: FUTURE-HIT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Siena (Other)
Collaborators: European Association of Cardiovascular Imaging (Other)
Responsible Party: Principal Investigator, Giulia Elena Mandoli, Principal Investigator, University of Siena
Other Study IDs: FUTURE_1.4
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mid Range Ejection Fraction; Heart Failure With Reduced Ejection Fraction
Keywords: Acute Heart Failure; Cronic Heart Failure; Progrostic Score; Transthoracic Echocardiography; Strain Echocardiography
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography — LV dimensions, LV mass and indices of LV function LA area and volume Indices of diastolic function (E/A ratio, E/e' ratio) Heart valve assessment according to GL RV dimensions and indices of RV function PAPs (RV-RA gradient and vena cava dimensions and collapsibility) B-lines at lung ultrasounds (comet lung score) Speckle Tracking analysis of LV (GLS), LA (PALS) and RV (LS of free wall) Optional 3D analysis of left and right ventricle

SUMMARY:
Acute heart failure (AHF) is defined as rapid onset or rapid worsening of typical signs and symptoms of heart failure (HF) according to the 2016 European Society of Cardiology Guidelines. AHF is the first cause of hospitalization in people over 65 in Western countries, accounting for more than 1 million hospitalizations per year in the USA. This disease has many repercussions not only in terms of mortality and morbidity, but also in terms of resources and infrastructures necessary for these patients' treatment, which constitutes a high economic burden for the national health care system. Even with growing knowledge and means, nowadays, the prognosis of AHF is still poor and there are no proven therapies that lead to long-term benefits in terms of reduced mortality. A better management of the acute phase of decompensation, including the definition of effective diagnostic-therapeutic workup and the use of innovative drugs, could improve the course of the disease, with positive effects on the patient (gain in survival and reduction of admissions), but also on the community (containment of the overall health costs). In recent years, numerous scores have been outlined in various AHF settings, considering only a small number of parameters. Several prognostic models have been developed suggesting how difficult it is to evaluate the AHF patients' prognosis. All this effort towards the development of so numerous prognostic models is justified by the fact that, despite the evolution of treatments, the risk of re-hospitalization and of both intrahospital mortality and after discharge remains high. Several studies have investigated potential prognostic factors that could help evaluating the risk of cardiovascular events, but now there is no accurate and complete prognostic score, particularly for AHF patients. Therefore, to date there are no accurate scores or determinants of short- and medium-term prognosis that allow to improve the management of these patients. This will be an observational, prospective, multicentric, international, non-commercial (non-profit) study. The primary endpoint will be to evaluate the best parameters, among clinical, laboratory and echocardiographic variables assessed within 24 hours from the hospital admission and before discharge, that are able to predict rehospitalization for HF and cardiovascular death at 3 and 6 months, in patients admitted to the cardiology department for acute exacerbation of chronic HF or de novo AHF.

DETAILED DESCRIPTION:
Acute heart failure (AHF), is defined as rapid onset or rapid worsening of typical signs and symptoms of heart failure (HF), according to the 2016 European Society of Cardiology Guidelines. It is a dangerous clinical condition for patient's life and requires urgent assessment and treatment, which typically lead to the patient's hospitalization. AHF is the first cause of hospitalization in people over 65 in Western countries, accounting for more than 1 million hospitalizations per year in the US. The one-year rehospitalization rate is higher among patients with acute onset of HF rather than among the ones with chronic HF (CHF) (30.7 vs 22.7). In cases of AHF, cardiovascular causes are responsible for readmission in 23.8% of the cases, whereas non-cardiovascular cases accounts for 8.3% of the cases. The rate of rehospitalization in de novo patients is lower than the one observed in subjects with known prior heart failure (8.2% vs 21.4%). In outpatients with CHF, the rehospitalization rate is roughly 22.7%, but only 8.8% is due to a new episode of HF. Our knowledge of the epidemiology of AHF is based primarily on various large-scale registries conducted both in the USA and in Europe. This disease has many repercussions not only in terms of mortality and morbidity, but also in terms of resources and infrastructures necessary for these patients' treatment, which constitutes a high economic burden for the national health care system. Even with growing knowledge and means, nowadays, the prognosis of AHF is still poor and there are no proven therapies that lead to long-term benefits in terms of reduced mortality. A better management of the acute phase of decompensation, including the definition of effective diagnostic-therapeutic workup and the use of innovative drugs, could improve the course of the disease, with positive effects on the patient (gain in survival and reduction of admissions), but also on the community (containment of the overall health costs). Several studies have investigated potential prognostic factors that could help evaluating the risk of cardiovascular events in HF patients, but now there is no accurate and complete prognostic score (that includes anamnestic, clinical, laboratory and echocardiographic parameters), particularly for AHF patients after their admission to the hospital. In recent years, numerous scores have been outlined in various AHF settings, considering only a small number of parameters. The role of echocardiography in the prognostic stratification of HF patients has been extensively studied. Several echocardiographic parameters have been evaluated, such as the dimensions of different cardiac chambers, the diastolic function of both the left (LV) and right ventricle (RV), and LV ejection fraction (LVEF). Several prognostic models have been developed, each of which uses a different combination of variables, suggesting how difficult it is to evaluate the AHF patients' prognosis. All this effort towards the development of so numerous prognostic models is justified by the fact that, despite the evolution of treatments, the risk of rehospitalization and of both intra-hospital mortality and after discharge remains high. LVEF is probably the most studied parameter and has been proven to be an important predictor of short-term and long-term mortality in AHF patients. LV compliance and filling pressures have also been extensively studied through traditional echocardiography. However, available data on the E/e' ratio and its prognostic value in patients with AHF is scarce and often conflicting, in fact some studies have shown that its lack of prognostic value, whereas others suggest that it can identify patients at higher risk of death and hospitalization, if combined to LVEF. Another important parameter to take into account is the systolic pulmonary arterial pressure (PAPs) which has been shown to be an important independent predictor of cardiovascular events. Recently, several studies have included new echocardiographic parameters in the evaluation of these patients' prognosis. Speckle Tracking Echocardiography (STE) is a non-invasive method that allows the assessment of the global and regional ventricular function of both the ventricles and the atria, independently of the angle of insonation. STE is based on the observation that the interaction between the ultrasound beam and the myocardium generates acoustic markers, defined speckle, which can be tracked in their displacement during the cardiac cycle, thanks to a dedicated software. The LV longitudinal strain (LS) represents the myocardial shortening along its longitudinal axis and it is identified by negative curves during systole and by positive ones in diastole. The LS is evaluated in 2-, 3- and 4-chamber apical views: global LS (GLS) is represented by the mean value of the deformation peak of the 18 obtained segments. LS of the RV (RVLS) is obtained in 4-chamber apical view and the segments of interest are 6 (3 for the free wall and 3 for the interventricular septum). Restricting the region of interest to the basal, middle and apical segments of RV free wall, it is possible to analyse the LS of this wall, leaving out the interventricular septum. STE has also been applied to the left atrium (LA) in order to assess its function. Two longitudinal strain parameters of the LA are recognized: the peak atrial LS (PALS), measured at the end of the atrial reservoir phase, and the peak atrial contraction strain (PACS), identified just before the start of the active atrial contraction. In recent years, the application of ultrasounds to the lungs has acquired relevance in the acute setting, in particular in determining the presence of congestion by the analysis of the so-called B lines. The latter represents comet artefacts that originate from the pleural line and they extend vertically towards the bottom of the screen, moving synchronously to the sliding of the lung during the breathing acts. Therefore, despite great effort, to date there are no accurate scores or determinants of short- and medium-term prognosis that allow to improve the management of these patients, keeping also in mind that this would allow the optimization of public spending. The FUTURE study population will prospectively recruit patients who will be admitted to a Coronary Intensive Care Unit or a cardiologic ward for AHF (including both acute exacerbation of chronic heart failure and first episode - de novo; the two populations will be also separately analysed). The basic statistical analysis will evaluate the demographic, clinical and echocardiographic parameters of the study population. The investigation will then focus on the identification of the parameters, among those that were collected, that at the end of the follow up period will be able to predict with greater sensitivity and specificity the risk of re-hospitalization and/or cardiovascular death at 3 and 6 months. A specific prognostic score will be then created from the obtained data, and its field of application would be all hospitalized patients for AHF, in order to predict the short- and medium- term outcome. Furthermore, a statistical sub-analysis will be performed to assess whether the selected prognostic parameters are valid even if the population is divided into 3 groups on the basis of LVEF (as indicated by the ESC guidelines, HFpEF, HFmrEF, HFpEF).

LV dimensions will be measured in parasternal long axis view. LV volumes, LA volume and area will be evaluated in 2- and 4- apical chamber view using the Simpson biplane method as indicated in the ASE recommendations. LV mass will be calculated from the 2D images with the trunk ellipsoid technique. The diastolic phase will be assessed through Pulsed-wave Doppler recordings of trans-mitral flow obtained from the apical 4-chamber view, by placing the sample volume at the level of the valve leaflet tips. Pulsed tissue Doppler imaging (TDI) will be used to measure annular velocities by placing the sample volume at the level of the lateral and septal angle of the mitral annulus from the apical 4-chamber view. Subsequently, the systolic (s'), early diastolic (e') and late (a') diastolic velocities will be obtained by averaging the values obtained. The E/e' ratio will be used as an index of the LV filling pressures. Mitral annulus plane systolic excursion will be assessed using Standard M-mode technique with the cursor placed at the lateral angle of the mitral annulus. From 4-chamber apical view, RV area will be measured both at the end of diastole and at the end of systole. The RV Fractional Area Change will be calculated. Mid-cavity RV linear dimension will be measured halfway between the maximal basal diameter and the apex, at the level of papillary muscles at end-diastole. Sphericity index of the RV will be evaluated as the ratio between the RV late-diastolic diameter and the RV longitudinal axis. RV longitudinal function will be assessed in apical 4-chamber view using TDI at the level of the lateral annulus of the tricuspid valve. The systolic peak velocity (s') will be used as an index of RV longitudinal function together with the tricuspid annulus plane systolic excursion evaluated in M-mode by placing the cursor at the lateral angle of the tricuspid annulus. 2D-STE will be performed from 4- and 2-chamber apical views of the conventional 2D gray-scale images, during a brief breath-hold and with a stable electrocardiographic trace. Particular attention should be paid to the acquisition of an adequate image that allows a clear discrimination of myocardial tissues and extra-cardiac structures. Three consecutive cardiac cycles will be recorded. The frame rate will be set between 40-80 frames/sec. The images acquired in this way will be processed using an appropriate software, with a semi-automatic method of analysing the strain based on the spatial motion of the speckles. The assessment of LV GLS, RV free wall LS and PALS will be performed in accordance to the ASE/EAE Consensus.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* admission to the cardiology departments for acute heart failure (de novo or exacerbation of chronic heart fail-ure) according to the clinical and instrumental criteria in the current ESC guidelines
* signing of the informed consent

Exclusion Criteria:

* age < 18 years
* valve prosthesis
* previous heart transplant or LVAD
* poor acoustic window.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The FUTURE study population will prospectively recruit patients who will be admitted to a Coronary Intensive Care Unit or a cardiologic ward for AHF (including both acute exacerbation of chronic heart failure and first episode - de novo; the two populations will be also separately analysed). Patients will be recruited at various centres around the world with no restrictions on ethnicity, etiology, LVEF value at the time of admission, and concomitant drug therapies. They will be selected exclusively on the basis of the authorization obtained through the signing of the informed consent and the presence of a good acoustic echocardiographic window.
Sampling Method: Non-Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
predictors of rehospitalization for heart failure and cardiovascular death | 3 and 6 months post discharge
  The primary endpoint of the FUTURE HIT study will be to evaluate the best parameters, among clinical, labora-tory and echocardiographic variables assessed within 24 hours from the hospital admission and before discharge, that are able to predict rehospitalization for HF and cardiovascular death at 3 and 6 months, in patients admitted to the cardiology department for acute exacerbation of CHF or de novo AHF.

SECONDARY OUTCOMES:
combined prognostic score of rehospitalization for heart failure and cardiovascular death | 3 and 6 months post discharge
  Creation of a combined prognostic dimensionsless score, using the parameters that came out as statistically significant towards the primary endpoint on a multicenter basis. Higher scores mean a worse outcome.
Event analysis according to heart failure's different classes (HFpEF, HFmrEF, HFrEF) | 3 and 6 months post discharge
  To analyze the events and the predictive ability of the parameters that came out as statistically significant to-wards the primary endpoint in the heart failure's different classes indicated in the guidelines (HFpEF, HFmrEF, HFrEF);
Event analysis according to genres | 3 and 6 months post discharge
  To analyze the events and predictive ability of the parameters in the two genres

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Cameli, Prof, Principal Investigator — Department of Medical Biotechnologies Division of Cardiology University of Siena
Locations (31):
- Blacktown Hospital, Faculty of Medicine, University of Sydney, Sydney, Australia
- Department of Cardiology, Antwerp University Hospital, Edegem, Belgium
- Greece (8):
  - Hygeia Hospital, Athens
  - Laiko General Hospital, Athens
  - Red Cross Hospital, Athens
  - General Hospital of Elefsina Thriassio, Elefsina
  - Onassis Cardiac Surgery center, Kallithea
  - Tzaneion General Hospital, Piraeus
  - 1st Cardiology Department, AHEPA University Hospital, Thessaloniki
  - Hippokrateion University Hospital, Medical School, Aristotle University of Thessaloniki, Third Cardiology Department, Thessaloniki
- Italy (12):
  - Centro Cardiologico Monzino IRCCS, Department of Cardiovascular Imaging, Milan
  - Division of Cardiology, Nephro-Cardiovascular Department, "S. Agostino- Estense" Public Hospital, University of Modena and Reggio Emilia, Modena
  - Division of Cardiology, A.O.R.N. "Sant'Anna e San Sebastiano", Caserta; Department of Translational Medical Sciences, University of Campania "Luigi Vanvitelli", Napoli
  - Federico II" University Hospital, Napoli
  - Dipartimento Toraco-Cardio-Vascolare, AOU Maggiore della Carità, Università del Piemonte Orientale, Novara
  - Cardiology Unit, Department of Excellence of Sciences for Health Promotion and Mothernal-Child Care, Internal Medicine and Specialities (ProMISE), University of Palermo, University Hospital Paolo Giaccone, Palermo
  - Unità Operativa di Cardiologia, Ospedale Guglielmo da Saliceto, Piacenza
  - Division of Cardiology; Department of Surgical, Medical and Molecular Pathology and Critical Care Medicine, AOUP, Pisa
  - Fondazione Toscana G. Monasterio, Pisa
  - Division of Cardiology - Nocera Inferiore Hospital and L. Vanvitelli University, Salerno
  - Heart Department, AOU S. Giovanni e Ruggi, Salerno, Italy., Salerno
  - Department of Medical Biotechnologies Division of Cardiology University of Siena, Siena
- National Institute of Cardiology of Mexico Ignacio Chávez, Mexico City, Mexico
- Department of Cardiology, Amsterdam University Medical Center, Amsterdam, Netherlands
- University Clinic- Department of Cardiology, St Cyril and Methodius University, R. of North Macedonia, Skopje, North Macedonia
- Centro Hospitalar Universitário de São João, Porto, Portugal
- Emergency Central Militar Hospital, Bucharest, Romania
- Hospital Vall d'Hebron, Barcelona, Spain
- Department of Cardiology, FSI Hospital, La Marsa, Tunisia
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Dr Siyami Ersek Cardiothoracic Surgery Center, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Eriksson H, Svardsudd K, Larsson B, Ohlson LO, Tibblin G, Welin L, Wilhelmsen L. Risk factors for heart failure in the general population: the study of men born in 1913. Eur Heart J. 1989 Jul;10(7):647-56. doi: 10.1093/oxfordjournals.eurheartj.a059542. PMID 2788575
- [Background] Cowie MR, Wood DA, Coats AJ, Thompson SG, Poole-Wilson PA, Suresh V, Sutton GC. Incidence and aetiology of heart failure; a population-based study. Eur Heart J. 1999 Mar;20(6):421-8. doi: 10.1053/euhj.1998.1280. PMID 10213345
- [Background] Guha K, McDonagh T. Heart failure epidemiology: European perspective. Curr Cardiol Rev. 2013 May;9(2):123-7. doi: 10.2174/1573403x11309020005. PMID 23597298
- [Background] Murphy NF, Simpson CR, McAlister FA, Stewart S, MacIntyre K, Kirkpatrick M, Chalmers J, Redpath A, Capewell S, McMurray JJ. National survey of the prevalence, incidence, primary care burden, and treatment of heart failure in Scotland. Heart. 2004 Oct;90(10):1129-36. doi: 10.1136/hrt.2003.029553. PMID 15367505
- [Background] Corrao G, Maggioni AP. [Epidemiology of heart failure]. G Ital Cardiol (Rome). 2014 Feb;15(2 Suppl 2):10S-15S. doi: 10.1714/1465.16183. Italian. PMID 24770484
- [Background] Tavazzi L, Senni M, Metra M, Gorini M, Cacciatore G, Chinaglia A, Di Lenarda A, Mortara A, Oliva F, Maggioni AP; IN-HF (Italian Network on Heart Failure) Outcome Investigators. Multicenter prospective observational study on acute and chronic heart failure: one-year follow-up results of IN-HF (Italian Network on Heart Failure) outcome registry. Circ Heart Fail. 2013 May;6(3):473-81. doi: 10.1161/CIRCHEARTFAILURE.112.000161. Epub 2013 Mar 8. PMID 23476054
- [Background] Kurmani S, Squire I. Acute Heart Failure: Definition, Classification and Epidemiology. Curr Heart Fail Rep. 2017 Oct;14(5):385-392. doi: 10.1007/s11897-017-0351-y. PMID 28785969
- [Background] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257
- [Background] O'Connor CM, Abraham WT, Albert NM, Clare R, Gattis Stough W, Gheorghiade M, Greenberg BH, Yancy CW, Young JB, Fonarow GC. Predictors of mortality after discharge in patients hospitalized with heart failure: an analysis from the Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF). Am Heart J. 2008 Oct;156(4):662-73. doi: 10.1016/j.ahj.2008.04.030. PMID 18926148
- [Background] Cleland JG, Swedberg K, Follath F, Komajda M, Cohen-Solal A, Aguilar JC, Dietz R, Gavazzi A, Hobbs R, Korewicki J, Madeira HC, Moiseyev VS, Preda I, van Gilst WH, Widimsky J, Freemantle N, Eastaugh J, Mason J; Study Group on Diagnosis of the Working Group on Heart Failure of the European Society of Cardiology. The EuroHeart Failure survey programme-- a survey on the quality of care among patients with heart failure in Europe. Part 1: patient characteristics and diagnosis. Eur Heart J. 2003 Mar;24(5):442-63. doi: 10.1016/s0195-668x(02)00823-0. PMID 12633546
- [Background] Komajda M, Follath F, Swedberg K, Cleland J, Aguilar JC, Cohen-Solal A, Dietz R, Gavazzi A, Van Gilst WH, Hobbs R, Korewicki J, Madeira HC, Moiseyev VS, Preda I, Widimsky J, Freemantle N, Eastaugh J, Mason J; Study Group on Diagnosis of the Working Group on Heart Failure of the European Society of Cardiology. The EuroHeart Failure Survey programme--a survey on the quality of care among patients with heart failure in Europe. Part 2: treatment. Eur Heart J. 2003 Mar;24(5):464-74. doi: 10.1016/s0195-668x(02)00700-5. PMID 12633547
- [Background] Maggioni AP, Dahlstrom U, Filippatos G, Chioncel O, Crespo Leiro M, Drozdz J, Fruhwald F, Gullestad L, Logeart D, Fabbri G, Urso R, Metra M, Parissis J, Persson H, Ponikowski P, Rauchhaus M, Voors AA, Nielsen OW, Zannad F, Tavazzi L; Heart Failure Association of the European Society of Cardiology (HFA). EURObservational Research Programme: regional differences and 1-year follow-up results of the Heart Failure Pilot Survey (ESC-HF Pilot). Eur J Heart Fail. 2013 Jul;15(7):808-17. doi: 10.1093/eurjhf/hft050. Epub 2013 Mar 28. PMID 23537547
- [Background] Follath F, Yilmaz MB, Delgado JF, Parissis JT, Porcher R, Gayat E, Burrows N, McLean A, Vilas-Boas F, Mebazaa A. Clinical presentation, management and outcomes in the Acute Heart Failure Global Survey of Standard Treatment (ALARM-HF). Intensive Care Med. 2011 Apr;37(4):619-26. doi: 10.1007/s00134-010-2113-0. Epub 2011 Jan 6. PMID 21210078
- [Background] Suzuki S, Yoshihisa A, Sato Y, Kanno Y, Watanabe S, Abe S, Sato T, Oikawa M, Kobayashi A, Yamaki T, Kunii H, Nakazato K, Ishida T, Takeishi Y. Clinical Significance of Get With the Guidelines-Heart Failure Risk Score in Patients With Chronic Heart Failure After Hospitalization. J Am Heart Assoc. 2018 Sep 4;7(17):e008316. doi: 10.1161/JAHA.117.008316. PMID 30371158
- [Background] Spinar J, Jarkovsky J, Spinarova L, Mebazaa A, Gayat E, Vitovec J, Linhart A, Widimsky P, Miklik R, Zeman K, Belohlavek J, Malek F, Felsoci M, Kettner J, Ostadal P, Cihalik C, Vaclavik J, Taborsky M, Dusek L, Littnerova S, Parenica J. AHEAD score--Long-term risk classification in acute heart failure. Int J Cardiol. 2016 Jan 1;202:21-6. doi: 10.1016/j.ijcard.2015.08.187. Epub 2015 Aug 28. PMID 26386914
- [Background] Magnussen C, Blankenberg S. Biomarkers for heart failure: small molecules with high clinical relevance. J Intern Med. 2018 Jun;283(6):530-543. doi: 10.1111/joim.12756. Epub 2018 Apr 22. PMID 29682806
- [Background] Soares FLJ, Oliveira JMG, Freire GNDC, Andrade LC, Noya-Rabelo MM, Correia LCL. Incremental Prognostic Value of Conventional Echocardiography in Patients with Acutely Decompensated Heart Failure. Arq Bras Cardiol. 2017 Dec;109(6):560-568. doi: 10.5935/abc.20170173. Epub 2017 Nov 27. PMID 29185616
- [Background] Adamopoulos C, Zannad F, Fay R, Mebazaa A, Cohen-Solal A, Guize L, Juilliere Y, Alla F. Ejection fraction and blood pressure are important and interactive predictors of 4-week mortality in severe acute heart failure. Eur J Heart Fail. 2007 Sep;9(9):935-41. doi: 10.1016/j.ejheart.2007.06.001. Epub 2007 Jul 12. PMID 17627880
- [Background] Hirata K, Hyodo E, Hozumi T, Kita R, Hirose M, Sakanoue Y, Nishida Y, Kawarabayashi T, Yoshiyama M, Yoshikawa J, Akasaka T. Usefulness of a combination of systolic function by left ventricular ejection fraction and diastolic function by E/E' to predict prognosis in patients with heart failure. Am J Cardiol. 2009 May 1;103(9):1275-9. doi: 10.1016/j.amjcard.2009.01.024. Epub 2009 Mar 9. PMID 19406271
- [Background] Wang M, Yip GW, Wang AY, Zhang Y, Ho PY, Tse MK, Lam PK, Sanderson JE. Peak early diastolic mitral annulus velocity by tissue Doppler imaging adds independent and incremental prognostic value. J Am Coll Cardiol. 2003 Mar 5;41(5):820-6. doi: 10.1016/s0735-1097(02)02921-2. PMID 12628728
- [Background] Shah RV, Chen-Tournoux AA, Picard MH, van Kimmenade RR, Januzzi JL. Galectin-3, cardiac structure and function, and long-term mortality in patients with acutely decompensated heart failure. Eur J Heart Fail. 2010 Aug;12(8):826-32. doi: 10.1093/eurjhf/hfq091. Epub 2010 Jun 5. PMID 20525986
- [Background] Arques S, Roux E, Ambrosi P, Sbragia P, Gelisse R, Pieri B, Luccioni R. Accuracy of bedside tissue Doppler echocardiography for the prediction of in-hospital mortality in elderly patients with acute heart failure with preserved left ventricular systolic function. comparison with B-type natriuretic peptide measurement. Int J Cardiol. 2007 Dec 15;123(1):69-72. doi: 10.1016/j.ijcard.2006.11.094. Epub 2007 Feb 6. PMID 17289178
- [Background] Aronson D, Darawsha W, Atamna A, Kaplan M, Makhoul BF, Mutlak D, Lessick J, Carasso S, Reisner S, Agmon Y, Dragu R, Azzam ZS. Pulmonary hypertension, right ventricular function, and clinical outcome in acute decompensated heart failure. J Card Fail. 2013 Oct;19(10):665-71. doi: 10.1016/j.cardfail.2013.08.007. PMID 24125104
- [Background] Merlos P, Nunez J, Sanchis J, Minana G, Palau P, Bodi V, Husser O, Santas E, Bondanza L, Chorro FJ. Echocardiographic estimation of pulmonary arterial systolic pressure in acute heart failure. Prognostic implications. Eur J Intern Med. 2013 Sep;24(6):562-7. doi: 10.1016/j.ejim.2013.04.009. Epub 2013 May 15. PMID 23684500
- [Background] Carluccio E, Dini FL, Biagioli P, Lauciello R, Simioniuc A, Zuchi C, Alunni G, Reboldi G, Marzilli M, Ambrosio G. The 'Echo Heart Failure Score': an echocardiographic risk prediction score of mortality in systolic heart failure. Eur J Heart Fail. 2013 Aug;15(8):868-76. doi: 10.1093/eurjhf/hft038. Epub 2013 Mar 19. PMID 23512095
- [Background] Cameli M, Mondillo S, Galderisi M, Mandoli GE, Ballo P, Nistri S, Capo V, D'Ascenzi F, D'Andrea A, Esposito R, Gallina S, Montisci R, Novo G, Rossi A, Mele D, Agricola E. [Speckle tracking echocardiography: a practical guide]. G Ital Cardiol (Rome). 2017 Apr;18(4):253-269. doi: 10.1714/2683.27469. Italian. PMID 28492566
- [Background] Mondillo S, Galderisi M, Mele D, Cameli M, Lomoriello VS, Zaca V, Ballo P, D'Andrea A, Muraru D, Losi M, Agricola E, D'Errico A, Buralli S, Sciomer S, Nistri S, Badano L; Echocardiography Study Group Of The Italian Society Of Cardiology (Rome, Italy). Speckle-tracking echocardiography: a new technique for assessing myocardial function. J Ultrasound Med. 2011 Jan;30(1):71-83. doi: 10.7863/jum.2011.30.1.71. PMID 21193707
- [Background] Meris A, Faletra F, Conca C, Klersy C, Regoli F, Klimusina J, Penco M, Pasotti E, Pedrazzini GB, Moccetti T, Auricchio A. Timing and magnitude of regional right ventricular function: a speckle tracking-derived strain study of normal subjects and patients with right ventricular dysfunction. J Am Soc Echocardiogr. 2010 Aug;23(8):823-31. doi: 10.1016/j.echo.2010.05.009. Epub 2010 Jun 19. PMID 20646910
- [Background] Cameli M, Caputo M, Mondillo S, Ballo P, Palmerini E, Lisi M, Marino E, Galderisi M. Feasibility and reference values of left atrial longitudinal strain imaging by two-dimensional speckle tracking. Cardiovasc Ultrasound. 2009 Feb 8;7:6. doi: 10.1186/1476-7120-7-6. PMID 19200402
- [Background] Cho GY, Marwick TH, Kim HS, Kim MK, Hong KS, Oh DJ. Global 2-dimensional strain as a new prognosticator in patients with heart failure. J Am Coll Cardiol. 2009 Aug 11;54(7):618-24. doi: 10.1016/j.jacc.2009.04.061. PMID 19660692
- [Background] Park JH, Park JJ, Park JB, Cho GY. Prognostic Value of Biventricular Strain in Risk Stratifying in Patients With Acute Heart Failure. J Am Heart Assoc. 2018 Oct 2;7(19):e009331. doi: 10.1161/JAHA.118.009331. PMID 30371332
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Jambrik Z, Monti S, Coppola V, Agricola E, Mottola G, Miniati M, Picano E. Usefulness of ultrasound lung comets as a nonradiologic sign of extravascular lung water. Am J Cardiol. 2004 May 15;93(10):1265-70. doi: 10.1016/j.amjcard.2004.02.012. PMID 15135701
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Quinones MA, Otto CM, Stoddard M, Waggoner A, Zoghbi WA; Doppler Quantification Task Force of the Nomenclature and Standards Committee of the American Society of Echocardiography. Recommendations for quantification of Doppler echocardiography: a report from the Doppler Quantification Task Force of the Nomenclature and Standards Committee of the American Society of Echocardiography. J Am Soc Echocardiogr. 2002 Feb;15(2):167-84. doi: 10.1067/mje.2002.120202. No abstract available. PMID 11836492
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Alexandru Popescu B, Waggoner AD; Houston, Texas; Oslo, Norway; Phoenix, Arizona; Nashville, Tennessee; Hamilton, Ontario, Canada; Uppsala, Sweden; Ghent and Liege, Belgium; Cleveland, Ohio; Novara, Italy; Rochester, Minnesota; Bucharest, Romania; and St. Louis, Missouri. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1321-1360. doi: 10.1093/ehjci/jew082. Epub 2016 Jul 15. No abstract available. PMID 27422899
- [Background] Mondillo S, Galderisi M, Ballo P, Marino PN; Study Group of Echocardiography of the Italian Society of Cardiology. Left ventricular systolic longitudinal function: comparison among simple M-mode, pulsed, and M-mode color tissue Doppler of mitral annulus in healthy individuals. J Am Soc Echocardiogr. 2006 Sep;19(9):1085-91. doi: 10.1016/j.echo.2006.04.005. PMID 16950462
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859